CLINICAL TRIAL: NCT02757573
Title: The Right Ventricular Responses to Mild Hypercarbia After Mitral Valve Repair Surgery - Assessment With Pulmonary Arterial Catheter and Transesophageal Echocardiography Measurements
Brief Title: The Right Ventricular Responses to Mild Hypercarbia After Mitral Valve Repair Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Kati Järvelä, MD, PhD, Tampere University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R16005
Record Dates: First submitted 2016-04-20; First posted 2016-05-02 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Heart; Decompensation, Right Ventricle; Echocardiography; Hypercapnia
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypercarbia (Experimental): Hypercarbia: PaCO2 is elevated from 5 to 7.5 kPa by controlled ventilation.
  Interventions: Procedure: Hypercarbia

INTERVENTIONS:
Procedure: Hypercarbia — PaCO2 is elevated from 5 to 7.5 kPa by controlled ventilation.

SUMMARY:
The aims of the study is to investigate the right ventricular responses to mild hypercarbia after mitral valve prolapse repair surgery by the measurements obtained on pulmonary arterial catheter and transesophageal echocardiography.

DETAILED DESCRIPTION:
The aims of the study is to investigate the right ventricular responses to mild hypercarbia after mitral valve prolapse repair surgery by the measurements obtained on pulmonary arterial catheter and transesophageal echocardiography. Investigators hypothesize that induced mild hypercarbia (PaCO2 7.5 kPa) cause elevated mean pulmonary arterial pressure and pulmonary vascular resistance, and this reflect to the right ventricle, both volume and function. And this right ventricle effect could be noticed by echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* scheduled mitral valve prolapse repair surgery
* able to give informed consent

Exclusion Criteria:

* preoperative right ventricular dysfunction or pulmonary hypertension
* significant tricuspid regurgitation
* congenital heart defect
* ventricular dyssynchrony or wide QRS-complex on ECG (> 130 ms)
* prior myocardial infarction (within tree months) or pericardial constriction
* preoperative left ventricular (LV) dysfunction, i.e. LV ejection fraction under 40 %
* if the scheduled repair by plastic procedure has been converted to mitral valve replacement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Tricuspid annular plane systolic excursion (TAPSE) | Change from baseline TAPSE at hypercarbia (in approximately 30 min)
  TAPSE will be measured at baseline (PaCO2 5 kPa) and at hypercarbia (PaCO2 7.5 kPa)
Mean pulmonary artery pressure (MPAP) | Change from baseline MPAP at hypercarbia (in approximately 30 min)
  MPAP will be measured at baseline (PaCO2 5 kPa) and at hypercarbia (PaCO2 7.5 kPa)

CONTACTS AND LOCATIONS:
Overall Officials: Kati Järvelä, MD, Principal Investigator — Tampere University Hospital; Kati Rautaneva, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital Heart Center, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tujunen MLJ, Lahti J, Kiiski H, Kuitunen AH, Tuohinen SS, Rautaneva K, Jalkanen VL, Huhtala H, Jarvela KM. Right Ventricular Response to Hypercapnia After Mitral Valve Repair: A Hemodynamic Assessment. Acta Anaesthesiol Scand. 2025 Jul;69(6):e70064. doi: 10.1111/aas.70064. PMID 40490845